CLINICAL TRIAL: NCT04294784
Title: A Multi-center, Open-label, Randomized Controlled Clinical Study of Nab-paclitaxel Plus SHR-1210(PD-1 Inhibitor)Versus Nab-paclitaxel As Second-line Treatment in Advanced or Recurrent Gastric and Esophagogastric Adenocarcinoma
Brief Title: Nab-paclitaxel Plus PD-1 Inhibitor Versus Nab-paclitaxel As Second-line Treatment in Advanced Gastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment forcing early suspension of screening and enrollment
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Head of the cancer center, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJCC011
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer
Keywords: Gastric cancer; GastroEsophageal Cancer; Albumin-bound Paclitaxel; PD-1 inhibitor
MeSH Terms: conditions — Stomach Neoplasms | interventions — Albumin-Bound Paclitaxel; camrelizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nab-P/PD-1 (Experimental): Patients in this arm receive albumin-bound paclitaxel and SHR-1210 (PD-1 inhibitor) thepary.
  Interventions: Drug: Albumin-bound Paclitaxel Plus SHR-1210 (PD-1 inhibitor)
- Nab-P (Active Comparator): Patients in this arm receive albumin-bound paclitaxel single-agent chemotherapy.
  Interventions: Drug: Albumin-bound Paclitaxel

INTERVENTIONS:
Drug: Albumin-bound Paclitaxel Plus SHR-1210 (PD-1 inhibitor) — Albumin-bound Paclitaxel 100 mg/m2,ivdrip,d1,d8,d15,Q28d,or Albumin-bound Paclitaxel 125-130 mg/m2,ivdrip,d1,d8,Q21d,or Albumin-bound Paclitaxel 260mg/m2,ivdrip,d1,Q21d;SHR-1210 200mg, ivdrip,d1,Q21d.
  Arms: Nab-P/PD-1
Drug: Albumin-bound Paclitaxel — Albumin-bound Paclitaxel 100 mg/m2,ivdrip,d1,d8,d15,Q28d,or Albumin-bound Paclitaxel 125-130 mg/m2,ivdrip,d1,d8,Q21d,or Albumin-bound Paclitaxel 260mg/m2,ivdrip,d1,Q21d;
  Arms: Nab-P

SUMMARY:
This is a Multi-center, Open-label, Randomized Controlled,phase 2 clinical trail of Albumin-bound Paclitaxel Plus SHR-1210 （PD-1 inhibitor）Versus Albumin-bound Paclitaxel as Second-line Treatment in Advanced or Recurrent Gastric Adenocarcinoma

DETAILED DESCRIPTION:
This is a Multi-center, Open-label, Randomized Controlled,phase 2 clinical trail of an immune checkpoint inhibitor in patients with advanced or recurrent gastric and esophagogastric junction adenocarcinoma, including two arms to compare the efficacy and safety of Albumin-bound Paclitaxel Plus SHR-1210 （PD-1 inhibitor）regimen and Albumin-bound Paclitaxel single-agent regimen in second-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-70 years.
2. Second line treatment for cytological or histological diagnosis of recurrent or metastatic gastric and esophagogastric adenocarcinoma. Disease progression after adjuvant therapy within 6 months is eligible.
3. ECOG performance status of 0-2.
4. Estimated life expectancy of at least 3 months.
5. Bone marrow function: white blood cell count≥3.0×109 /L, absolute neutrophil count(ANC) ≥1.5×109 /L, platelet count(PLT) ≥90×109 /L, hemoglobin(HB) ≥90 g/L.
6. Left ventricular ejection fraction (LVEF) ≥ 50%.
7. Liver and kidney function: Creatinine(Cr)≤1.5 x upper limit of normal range(ULN); alanine glutamate transaminase (ALT) and glutamate transaminase (AST) ≤2.5 x upper limit of normal range (ULN), or ≤5 x upper limit of normal range (ULN)when with hepatic metastases，total bilirubin (TBIL)≤1.5 x upper limit of normal range (ULN), or≤2.5 x upper limit of normal range (ULN) when with Gilbert's syndrome.
8. Any acute, clinically significant treatment-related toxicity caused by previous treatment must have been reduced to less than or equal to grade 1, except hair loss.
9. Able and willing to comply with the study plans in this protocol and sign the informed consent.

Exclusion Criteria:

1. uncontrollable infections or have received systematic antibiotic treatment within 72 hours before enrollment.
2. Any abnormal bone marrow hyperplasia or other abnormal hematopoietic function.
3. Have a second malignancy within 5 years prior to registration except for cured carcinoma in situ of cervix uteri, non-melanoma skin cancer.
4. Patients with symptomatic brain metastases.
5. Allergic to the chemotherapy drugs or the materials in this study.
6. Suffering from mental or nervous system disorders and unable to cooperate.
7. Pregnant or nursing female patients. Men and women of reproductive age are unwilling to take reliable contraceptive measures during the study.
8. Active autoimmune disease, history of autoimmune disease, use of corticosteroids or immunosuppressants, or use of hormone replacement therapy, such as thyroxine, insulin, etc.
9. Live vaccine was administered within 30 days before enrolment (injectable seasonal influenza vaccine is allowed as it is inactivated).
10. Patients with other diseases not suitable for enrolment, such as active tuberculosis, hepatitis B (after treatment, hepatitis B virus titer HBV-DNA <500IU/ml, and liver function is normal, but cannot be combined with hepatitis C), hepatitis C, uncontrolled electrolyte disorders ,pericardial effusion, pleural effusion and abdominal effusion, etc.
11. Have participated in other clinical trials within 30 days prior to this study.
12. History of organ transplantation.
13. Patients that researcher consider cannot sign informed consent or complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
objective response rate(ORR) | up to 12 months
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).Higher rate of ORR indicates better treatment effect.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 9 months
  Time from the start of treatment to progression of disease or death.Higher rate of 9m PFS in statistic analysis means better outcome.
Overall survival (OS) | up to 12 months
  Time from the start of treatment until death due to any reason.Increased rate of 12m OS compared to the other arm indicates more benefit from the treatment regimen.
Safety as measured by number and grade of adverse events | up to 12 months
  Summary adverse events according to NCI-CTCAE 5.0
patient-reported outcomes (PROs) | up to 12 months
  Patient-reported outcomes according to EQ-5D questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, MD,PhD, Study Chair — oncology center of Tongji Hospital,wuhan,China
Locations (1):
- Tongji hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun L, Gong Z, Wang L, Kuang L, Huang Q, Pei B, Yuan X, Qiu H. Multi-center phase II study of nab-paclitaxel plus camrelizumab versus nab-paclitaxel alone as second-line treatment for advanced gastric cancer. Oncologist. 2025 Jul 4;30(7):oyaf189. doi: 10.1093/oncolo/oyaf189. PMID 40554667